CLINICAL TRIAL: NCT01926912
Title: HOSPItal Use of Paliperidone Palmitate - A Prospective Non-Interventional Study
Brief Title: A Study of Usage of Paliperidone Palmitate in Patients With Schizophrenia in a Hospital Setting
Acronym: HOSPIPalm
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Other Study IDs: CR100862; R092670SCH4017 (Other: Janssen-Cilag International NV)
Record Dates: First submitted 2013-08-19; First posted 2013-08-21 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-08

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Paliperidone Palmitate; Hospital setting; Schizophrenic Disorders
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants with schizophrenia
  Interventions: Drug: No intervention

INTERVENTIONS:
Drug: No intervention — This is an observational study. Participants prescribed with paliperidone palmitate by the treating physician as per local labeling information in the hospital setting will be observed and data will be collected.

SUMMARY:
The purpose of this study to evaluate safety, tolerability, treatment outcomes, appropriate use and pattern of paliperidone palmitate usage in participants with schizophrenia in the hospital setting.

DETAILED DESCRIPTION:
This is a prospective (look forward using periodic observations collected predominantly following patient enrollment), multicenter, observational study (a type of study in which participants are observed or certain outcomes are measured). This study will consist of 6-week observational period during which data will be collected for participants who are hospitalized due to schizophrenia exacerbation and are receiving treatment with paliperidone palmitate (treatment initiated within 3 weeks after admission to hospital). The participant satisfaction will be evaluated at week 6 (or early discontinuation). Safety evaluations will include body weight, extrapyramidal symptom (eg, inability to initiate movement and inability to remain motionless) rating scale scores, concomitant therapy and assessment of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with schizophrenia
* Participant admitted to hospital due to an exacerbation of their schizophrenia prior to any study-related activity
* Participant may, in the opinion of the participating physician, benefit from treatment with paliperidone palmitate which will be initiated within 3 weeks after admission to hospital

Exclusion Criteria:

* Participant has a known hypersensitivity to paliperidone or risperidone
* Participant has previously been treated with paliperidone palmitate
* Participant has a history of neuroleptic malignant syndrome
* Participant was on clozapine or has previously been treated with any long-acting injectable antipsychotic during the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with schizophrenia receiving paliperidone palmitate in the hospital setting
Sampling Method: Non-Probability Sample
Enrollment: 371 (Actual)
Dates: Start 2013-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | Up to 6 weeks
Number of participants who discontinue the study due to adverse events | Up to 6 weeks

SECONDARY OUTCOMES:
Change from baseline in Extrapyramidal Symptom Rating Scale (ESRS) score | Baseline, Week 1, Week 2, Week 5, and Week 6
  The ESRS is a 12 item clinician-rated scale designed to assess the severety of extrapyramidal symptoms. Dyskinesic movements are rated according to bothfrequency and amplitude. It measures the four types of drug-induced movement disorders. (Parkinsonism, Dystonia, akathisia, and Dyskinesia). Items are rated on a 7-point scale ranging from 0 (normal) to 6 (extremely severe). The higher the score, the more severely the symptoms affect function. Higher scores indicate worsening.
Change from baseline in total Brief Psychiatric Rating Scale (BPRS) score | Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, and Week 6
  The BPRS is used for the measurement of psychiatric symptoms. The BPRS is an 18 item questionnaire and each question is rated on a 7 point scale ranging from 1 (not present) to 7 (extremely severe). The total score for the 18 question will be calculated by adding score of each question. The interpretation of the total scores are: 0-9 will indicate "not a schizoaffective case"; 10-20 will indicate "possible schizoaffective case"; and 21 or more, will indicate "evident schizoaffective case". Higher scores indicate worsening.
Clinical Global Impression - Severity (CGI-S) scale score | Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, and Week 6
  The CGI-S rating scale is a 7-point global assessment that measures the clinician's impression of the severity of illness exhibited by a participant. A rating of 1 is equivalent to "Normal, not at all ill" and a rating of 7 is equivalent to "Among the most extremely ill participants". Higher scores indicate worsening.
Clinical Global Impression - Change (CGI-C) scale score | Week 6
  The CGI-C is a 7-point assessment scale of change in global clinical status, defined as a sense of well-being and ability to function in daily activities. CGI-C scores range from 1 (very much improved) through to 7 (very much worse). Higher scores indicate worsening.
Change from baseline in Personal and Psychosocial functioning (PSP) scale score | Baseline and Week 6
  The PSP is used as a measure of personal and social functioning of participants with psychiatric disorders. The PSP scale assesses the degree of difficulty a participant exhibits over a 1-month period within 4 domains of behavior: socially useful activities, personal and social relationships, self-care, and disturbing and aggressive behavior and provide rating from 1 to 100. Participants with score of 71 to 100 have a mild degree of difficulty; from 31 to 70 have marked difficulty and from 1 to 30, have represent severe degrees of difficulty. Lower scores indicate worsening.
Subject Satisfaction with previous antipsychotic medication (MSQ) scale score | Baseline
  Treatment satisfaction with previous anti psychiatric medication among participants with schizophrenia will be assessed by using the MSQ scale. It consists of 1 question: "Overall, how satisfied are you with your current antipsychotic medication(s)?" with responses assessed on a 7-point scale rated as follows: 1=extremely dissatisfied, 2=very dissatisfied, 3=somewhat dissatisfied, 4=neither satisfied nor dissatisfied, 5=somewhat satisfied, 6=very satisfied, and 7=extremely satisfied. Lower scores indicate worsening.
Subject Satisfaction with study medication (paliperidone palmitate) scale score | Week 6
  Treatment satisfaction with study medication (paliperidone palmitate) among participants with schizophrenia will be assessed by using the MSQ scale. It consists of 1 question: "Overall, how satisfied are you with your current antipsychotic medication(s)?" with responses assessed on a 7-point scale rated as follows: 1=extremely dissatisfied, 2=very dissatisfied, 3=somewhat dissatisfied, 4=neither satisfied nor dissatisfied, 5=somewhat satisfied, 6=very satisfied, and 7=extremely satisfied. Lower scores indicate worsening.
Change from baseline in body weight | Baseline and Week 6

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (39):
- Belgium (3):
  - Diest
  - Saint-Servais
  - Tournai
- Bulgaria (6):
  - Pazardzhik
  - Rousse
  - Sofia
  - Stara Zagora
  - Targovishte
  - Vratsa
- Denmark (2):
  - Elsinore
  - København S
- Germany (9):
  - Berlin
  - Chemnitz
  - Dresden
  - Greifswald
  - Hamburg
  - Hennigsdorf
  - Neuruppin
  - Pfaffenhofen
  - Sachsen
- Greece (4):
  - Heraklion Crete
  - Ioannina
  - Katerini Pieria
  - Thessaloniki
- Israel (2):
  - Bat Yam
  - Tel Litwinsky
- Kazakhstan (5):
  - Almaty
  - Astana
  - Kyzylorda
  - Taraz
  - Ust-Kamenogorsk
- Russia (8):
  - Chelyabinsk
  - Moscow
  - Nizhny Novgorod
  - Omsk
  - Orenburg, Staritsa Village
  - Saint Petersburg
  - Tula Region
  - Yaroslavl

REFERENCES:
- See also: HOSPItal Use of Paliperidone Palmitate - A Prospective Non-Interventional Study — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=3530&filename=CR100862_CSR.pdf